CLINICAL TRIAL: NCT07002112
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of the LVIVO-TaVec100 Product in the Treatment of Relapsed/Refractory B-cell Malignancies
Brief Title: The LVIVO-TaVec100 Product in the Treatment of Relapsed/Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Principal Investigator, Lei Fan, Director of lymphoma center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2409-0001
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LVIVO-TaVec100 product (Experimental): Each subject will be given a single-dose LVIVO-TaVec100 product infusion at each dose level.
  Interventions: Biological: LVIVO-TaVec100 product

INTERVENTIONS:
Biological: LVIVO-TaVec100 product — Prior to infusion of the LVIVO-TaVec100 product, subjects will receive bridging therapy if needed.

SUMMARY:
A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of the LVIVO-TaVec100 product in the Treatment of Relapsed/Refractory B-cell Malignancies.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation/dose extension study to assess the safety, tolerability, and efficacy of LVIVO-TaVec100 product in the patient ≥ 18 years of age with relapsed or refractory B-cell Malignancies. Subjects who meet the eligibility criteria will receive a single dose of LVIVO-TaVec100 product. The study will include the following sequential phases: screening, bridging therapy (if needed), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical studies; Fully informed of this study and signed informed consent; Informed consent form must be obtained prior to initiation of any study-related tests or procedures that are not part of the standard treatment for the subject's disease; Good compliance and cooperation with follow-up.
2. Aged 18-65 years (inclusive).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. At least one evaluable tumor lesion.
5. Relapsed and/or refractory NHL , and relapsed and/or refractory CLL with treatment indications
6. Life expectancy≥ 3 months
7. Clinical laboratory values meet screening visit criteria
8. Adequate organ function;

Exclusion Criteria:

Subject eligible for this study must not meet any of the following criteria:

1. Prior antitumor therapy with insufficient washout period ;
2. Prior treatment with other autologous cells or gene therapies other than targeting CD19 autologous CAR-T;
3. Patients who are positive for hepatitis B surface antigen (HBsAg), hepatitis B virus core antibody (HBcAb), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), and human immunodeficiency virus antibody (HIV-Ab).
4. Known life-threatening allergic reaction, hypersensitivity reaction, or intolerance to study drug excipients and related excipients, including but not limited to DMSO; or those with a history of severe allergic reactions in the past (such as hypersensitivity reactions, or those with severe immune-related reactions such as the need for glucocorticoids to prevent anaphylaxis as assessed by the investigator).
5. Lactating women;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and type of TEAEs (Treatment-emergent Adverse Events) | Through study completion, an average of 2 years after LVIVO-TaVec100 infusion (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Pharmacokinetics in peripheral blood | Through study completion, an average of 2 years after LVIVO-TaVec100 infusion (Day 1)
  CAR positive T cells and CAR transgene percentage of in peripheral blood after LVIVO-TaVec100 infusion.
Pharmacokinetics in bone marrow | Through study completion, an average of 2 years after LVIVO-TaVec100 infusion (Day 1)
  CAR positive T cells and CAR transgene percentage of in bone marrow after LVIVO-TaVec100 infusion.
The recommended Phase II dose (RP2D) for this cell therapy | 30 days after LVIVO-TaVec100 infusion
  RP2D established through 3+3 design and the DLTs occurring following LVIVO-TaVec100 infusion

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average 2 years after LVIVO-TaVec100 infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LVIVO-TaVec100 cell infusion
Progression-free survival (PFS) | Through study completion, an average 2 years after LVIVO-TaVec100 infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LVIVO-TaVec100 to the first documented disease progression or death, whichever occurs first
Overall Survival (OS) | Through study completion, an average 2 years after LVIVO-TaVec100 infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LVIVO-TaVec100 to death of the subject
Time to Response (TTR) | Through study completion, an average 2 years after LVIVO-TaVec100 infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LVIVO-TaVec100 to the date of the first response evaluation of the subject who has met all criteria for CR or PR
Duration of Response (DoR) | Through study completion, an average 2 years after LVIVO-TaVec100 infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or PR) to the first documented relapse evidence of the responders
Immunogenicity assessment of LVIVO-TaVec100 infusion | Through study completion, an average 2 years after LVIVO-TaVec100 infusion (Day 1)
  The incidence of Anti- LVIVO-TaVec100 antibody in patients who received LVIVO-TaVec100 infusion

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of USTC west district, Hefei, Anhui
  - Beijing Gobroad Boren Hospita, Beijing, Beijing Municipality
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of ZHENGZHOU University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No